CLINICAL TRIAL: NCT04006587
Title: Incentive Spirometer Device Reduces Pulmonary Complications in Patients With Traumatic Rib Fractures
Brief Title: IS Reduces Rib Fracture Complications
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: CMRPG 2E0221
Record Dates: First submitted 2019-06-27; First posted 2019-07-05 (Actual); Last update posted 2019-07-05 (Actual); Status verified 2019-06

CONDITIONS: Hemothorax; Traumatic; Rib Fractures; Rib Trauma
Keywords: incentive spirometer; Hemothorax; Traumatic; trauma; rib Fractures
MeSH Terms: conditions — Hemothorax; Rib Fractures; Wounds and Injuries

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- IS intervention (Experimental): patients were instructed how to use the IS in a seated or semi-seated position, and to maintain sustained maximal inspiration for 3-5 seconds before exhalation, ten times per hour, and for at least eight hours a day.
  Interventions: Device: incentive spirometer
- control (No Intervention): standard care without IS intervention

INTERVENTIONS:
Device: incentive spirometer — patients were instructed how to use the IS in a seated or semi-seated position, and to maintain sustained maximal inspiration for 3-5 seconds before exhalation, ten times per hour, and for at least eight hours a day.
  Arms: IS intervention

SUMMARY:
The incentive spirometer (IS) is a mechanical device that helps lung expansion. It is commonly used to prevent postoperative lung atelectasis and decreased pulmonary complications in patients who received cardiac, lung, or abdomen surgery.This study aimed to explore the effect of the IS on the improvement of lung function and decrease in pulmonary complication rate in rib fractures patients.

DETAILED DESCRIPTION:
Adult patients (>18 years old) seen at our institution between June, 2014 until May, 2017 with traumatic rib fractures were included. For inclusion, a patient had to have at least one rib fracture as detected by chest X-ray (CXR) or computed tomography scan. We excluded patients with unconsciousness, history of chronic obstructive pulmonary disease, asthma, or an Injury Severity Score (ISS) ≥ 16. Patients were divided into two groups using a randomized envelope technique: in the study group, patients were advised to use the IS and in the control group patients did not received the IS. All patients were managed with the same oral analgesic protocol. A CXR was obtained on the 1st and 5th day of admission and performed by a radiologist. The Pulmonary Function Test (PFT) was administered on the 2nd and 7th day of admission and performed by a pulmonologist. A numeric rating scale (NRS) was used to define the severity of chest pain on the 1st and 5th day of admission.

ELIGIBILITY:
Inclusion Criteria:

* at least one rib fracture as detected by chest X-ray (CXR) or computed tomography scan

Exclusion Criteria:

* unconsciousness,
* history of chronic obstructive pulmonary disease
* asthma
* Injury Severity Score (ISS) ≥ 16

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2014-06-01 (Actual); Primary Completion 2017-05-31 (Actual); Study Completion 2017-06-01 (Actual)

PRIMARY OUTCOMES:
pulmonary complication rate | 2 weeks after trauma
  atelectasis, pneumonia, hemothorax, and pneumothorax

SECONDARY OUTCOMES:
1st lung function test | 2nd day of admission
  forced vital capacity and forced expiratory volume in 1 second
2nd lung function test | 7th day of admission
  forced vital capacity and forced expiratory volume in 1 second
length of hospital stay | total hospital stay days up to 2 months after admission
  total stay in hospital after trauma
1st Pain score | 1st day of admission
  Numerical Pain Rating Scale of chest pain, from 0 (no pain) to 10 (worst pain)
2nd Pain score | 5th day of admission
  Numerical Pain Rating Scale of chest pain, from 0 (no pain) to 10 (worst pain)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sum SK, Peng YC, Yin SY, Huang PF, Wang YC, Chen TP, Tung HH, Yeh CH. Using an incentive spirometer reduces pulmonary complications in patients with traumatic rib fractures: a randomized controlled trial. Trials. 2019 Dec 30;20(1):797. doi: 10.1186/s13063-019-3943-x. PMID 31888765